CLINICAL TRIAL: NCT03768739
Title: Dysphagia and Vocal Fold Mobility Impairment in Cardiac Surgical Patients
Brief Title: Dysphagia and VFMI in Cardiac Patients
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201802740
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Cardiac Disease
Keywords: Dysphagia; Extubation; Cardiac Intensive Care Unit (CICU); Forced Expiratory Volume in One second (FEV1); Peak Expiratory Flow (PEF)
MeSH Terms: conditions — Heart Diseases; Deglutition Disorders | interventions — Fees and Charges

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CICU extubated patients: Participants will undergo a Fiberoptic Endoscopic Evaluation of Swallowing (FEES)
  Interventions: Procedure: Fiberoptic Endoscopic Evaluation of Swallowing

INTERVENTIONS:
Procedure: Fiberoptic Endoscopic Evaluation of Swallowing — This procedure involves a flexible laryngoscope that contains a light source and video camera on the end through the open passages of your nose and to the back of the throat in order to visualize the swallowing mechanism.
  Other Names: FEES

SUMMARY:
The proposed study seeks to determine the incidence of dysphagia and vocal fold mobility impairment (VFMI) in individuals undergoing cardiothoracic surgical procedures. It also seeks to determine the impact of postoperative swallowing impairment on health-related outcomes.

DETAILED DESCRIPTION:
Swallowing impairment and VFMI are common, yet often overlooked, complications of cardiac surgical procedures. The true incidence of both dysphagia and VFMI in this patient population is unclear due to a lack of rigorous study using instrumental assessment techniques and validated outcomes in all patents undergoing cardiac surgery. We therefore aimed to determine the incidence of dysphagia and VFMI in this patient population and to characterize impairment profiles related to swallowing safety and efficiency. We also aimed to assess the relative impact of VFMI and dysphagia on health-related outcomes such as length of hospital stay, pneumonia, sepsis, reintubation, and discharge status.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 - 90 years old
* undergoing planned or emergent cardiothoracic surgery via sternotomy and/or extended thoracotomy requiring cardiopulmonary bypass
* willing to participate in post-operative swallowing evaluation testing

Exclusion Criteria:

* Patients undergoing exclusively transcatheter valves
* Patients undergoing exclusively thoracic endovascular aortic repair procedures
* The inability to achieve appropriate alertness and cognitive status following procedure will exclude one from completing the study.
* Participants must pass cognition, respiratory and physical abilities screening to ensure testing safety.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 230 individuals undergoing cardiothoracic surgery will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2019-02-03 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

PRIMARY OUTCOMES:
Penetration Aspiration Scale | Baseline
  This scale is a validated measure used by trained blinded clinicians to assign ratings of safety to swallowing bolus trials. The development and use of an 8-point, equal-appearing interval scale (8 being best; 1 being worst) to describe penetration and aspiration events are described. Scores are determined primarily by the depth to which material passes in the airway and by whether or not material entering the airway is expelled.
Yale Residue Severity Rating Scale | Baseline; Day 30
  This scale is a validated measure used by trained blinded clinicians to assign ratings of efficiency to swallowing bolus trials. The Yale Pharyngeal Residue Severity Rating Scale was developed, standardized, and validated to provide reliable, anatomically defined, and image-based assessment of post-swallow pharyngeal residue severity as observed during fiberoptic endoscopic evaluation of swallowing (FEES). It is a five-point ordinal rating scale based on residue location (vallecula and pyriform sinus) and amount (none, trace, mild, moderate, and severe)
Vocal Fold Mobility Impairment | Baseline
  Index of left and right vocal fold movement

CONTACTS AND LOCATIONS:
Overall Officials: Emily Plowman, PhD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - Cardiovascular Clinic at UF Health UF, Gainesville, Florida
  - UF Health at the University of Florida, Gainesville, Florida
  - Thoracic and Cardiovasscular Surgery at UF Health, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Plowman EK, Anderson A, York JD, DiBiase L, Vasilopoulos T, Arnaoutakis G, Beaver T, Martin T, Jeng EI. Dysphagia after cardiac surgery: Prevalence, risk factors, and associated outcomes. J Thorac Cardiovasc Surg. 2023 Feb;165(2):737-746.e3. doi: 10.1016/j.jtcvs.2021.02.087. Epub 2021 Mar 3. PMID 33814177